CLINICAL TRIAL: NCT01333163
Title: GLP-1: Acute Effects on Kidney Function in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeppe Skov (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Jeppe Skov, MD, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: VEKRM 29414
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Kidney Functional
MeSH Terms: interventions — Amides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 (Active Comparator)
  Interventions: Biological: Human GLP-1 (7-36) amide
- Placebo (Placebo Comparator)
  Interventions: Biological: Isotone NaCl

INTERVENTIONS:
Biological: Human GLP-1 (7-36) amide — 2 hour IV infusion, 1,5pmol/min/kg.
  Arms: GLP-1
Biological: Isotone NaCl — 2 hours IV infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate how Glucagon-Like Peptide 1 (GLP-1) affects kidney function in healthy young men. The hypothesis is that GLP-1 induces a positive effect on kidney hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men

Exclusion Criteria:

* Any chronic diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | Every 20 minutes for 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Skov, MD, Principal Investigator — University of Aarhus
Locations (1):
- Klinisk Institut, Afd. MEA, Aarhus Sygehus, NBG, Aarhus C, Denmark

REFERENCES:
- [Derived] Skov J, Dejgaard A, Frokiaer J, Holst JJ, Jonassen T, Rittig S, Christiansen JS. Glucagon-like peptide-1 (GLP-1): effect on kidney hemodynamics and renin-angiotensin-aldosterone system in healthy men. J Clin Endocrinol Metab. 2013 Apr;98(4):E664-71. doi: 10.1210/jc.2012-3855. Epub 2013 Mar 5. PMID 23463656